CLINICAL TRIAL: NCT06254183
Title: Clinical Study Evaluating the Effect of Gabapentin on Kidney Function Following Laparoscopic Sleeve Gastrectomy (LSG) for Morbid Obese Patients
Brief Title: Effect of Gabapentin on Kidney Function Following Laparoscopic Sleeve Gastrectomy(LSG)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Kholoud Salah Ibrahim Amin, Principle Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Gabapentin use in LSG
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury; Bariatric Surgery Candidate; Gabapentin
MeSH Terms: conditions — Acute Kidney Injury | interventions — Gabapentin; gamma-Aminobutyric Acid

STUDY DESIGN:
Intervention Model Description: Group I: 30 patients who will represent the control group and will receive oral placebo tab 2 days prior to surgery and 1 hr before surgery.
  Group II: 30 patients who will represent the treatment group and will receive a single oral dose of Gabapentin 1200 mg, 1 hr before surgery.
  Blood and urine samples will be collected before the surgery, then 24 hrs postoperatively.
  Blood and urine samples will be collected in follow-up, 6 months postoperatively
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Active Comparator): 30 patients will represent the treatment group and will receive a single oral dose of Gabapentin 1200 mg 1 hr before the surgery.
  Blood and urine samples will be collected before the surgery, then 24 hrs postoperatively.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): 30 patients will represent the treatment group and will receive a single oral dose of Placebo 1 hr before the surgery.
  Blood and urine samples will be collected before the surgery, then 24 hrs postoperatively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin is a drug that is commonly used to treat neuropathic pain, epilepsy, and other neurological disorders. According to some studies, gabapentin may affect the Wnt signaling pathway.
  In this study Gabapentin will be given by a dose of 1200 mg 1 hour before a laparoscopic sleeve gastrectomy(LSG) to decrease postoperative pain and opioid consumption. As acute kidney injury is a common condition following LSG , and as gabapentin has a positive effect on decreasing AKI induced in animal studies, we assess the effect of gabapentin on the AKI status following LSG
  Other Names: GABA
  Arms: Gabapentin
Drug: Placebo — A placebo is a sham medical treatment that appears to be a real medical intervention but has no therapeutic effect. It is often used in clinical trials to compare the effects of a new treatment to those of a placebo. Common examples of placebos include inert tablets (like sugar pills), inert injections (like saline), and even sham surgery or other procedures. Placebos are typically made of inactive substances such as starch or sugar and are designed to be indistinguishable from the actual treatment
  Arms: Placebo

SUMMARY:
Assessment of the effect of gabapentin as an analgesic replacement on the Kidney function following Laparoscopic sleeve gastrectomy for Morbid Obese Patients by measuring two biomarkers: NGAL (Neutrophil gelatinase-associated lipocalin)and DKK3 (Dickkopf-3)

DETAILED DESCRIPTION:
Obesity should be viewed as the number one preventable risk factor for kidney disease because obesity mediates the majority of diabetes and hypertension, the 2 major causes of end-stage kidney disease (ESKD). Morbidly obese adults have a 6-fold higher risk of diabetes compared with their lean peers.

Laparoscopic sleeve gastrectomy (LSG) has been approved since 2010, by both the American Society for Metabolic and Bariatric Surgery (ASMBS) and the American College of Surgeons (ACS) as an operation for the treatment of obesity and other obesity-related diseases.

Acute kidney injury (AKI) is one of the most common postoperative complications. It is a serious morbidity occurring during hospitalizations, and it is associated with prolonged hospital stay, high risk of in-hospital mortality, increased hospital costs, and decreased survival for up to 15 years after surgery. In addition, AKI increases the risk of incident and progressive chronic kidney disease and is associated with reduced long-term survival.

Non-steroidal anti-inflammatory drugs (NSAIDs) represent one of the most common classes of medications used postoperatively. It is estimated that 1-5% of NSAIDs users may develop renal adverse effects, both AKI and CKD.

Gabapentin, an anticonvulsant widely used for the treatment of various neuropathic pain syndromes, has recently been investigated as an analgesic agent in the perioperative setting. Although it is not an analgesic itself, early experience suggests this medication can improve pain and reduce opioid requirements.

A new animal study shows that gabapentin demonstrated reno-protective properties against either acute or chronic kidney injury, primarily attributed to its antioxidant properties. Further clinical studies are required to validate and standardize therapeutic doses of gabapentin under investigation in patients susceptible or at risk of developing kidney dysfunction.

In this study, Neutrophil gelatinase-associated lipocalin (NGAL) and Dickkopf-3 (DKK3) will be biomarkers to assess kidney function. NGAL appears to be a promising marker for early detection of AKI and is likely to be adapted for wide-scale clinical use in patient management as a point-of-care test.

Measurement of DKK3 in urine represents a novel tool for the identification of patients at high risk for AKI regardless of the cause of kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese patients with normal kidney function, undergoing Laparoscopic sleeve gastrectomy surgery.
* Both sexes.
* Age ≥ 18 years

Exclusion Criteria:

* • Patients have advanced cancer on active treatment and end-stage renal, hepatic, and cardiopulmonary disease.

  * Patients with untreated schizophrenia, cognitive impairment and using psychiatric medications.
  * Patients with active substance abuse.
  * Patients on chronic dosage of Gabapentin or allergic to it.
  * Pregnant women or women on breastfeeding.
  * Patients on medications that could interfere with assessed parameters will be excluded.

The ethical approval of the study will be obtained from by Medical research Ethics Committee of Tanta and Mansoura Universities and all participants will give their written consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Level of Neutrophil gelatinase-associated lipocalin (NGAL) | up to 6 months postoperative
  Neutrophil gelatinase-associated lipocalin in Serum using ELISA Kits
Level of Dickkopf-3 (DKK3) | up to 6 months postoperative
  Dickkopf-3 in both serum and urine using ELISA kits

SECONDARY OUTCOMES:
Kidney function test | up to 6 months postoperative
  Blood urea nitrogen
level of Serum creatinine | up to 6 months postoperative
lipid profile (Triglycerides, LDL, HDL) | up to 6 months postoperative
Concentration of calcium in serum | up to 6 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Kamal Tawfeek Hegazy, Professor, Principal Investigator — Tanta University; Ahmed Mohammed Hassan Shata, Professor, Study Director — Mansoura University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kovesdy CP, Furth SL, Zoccali C; World Kidney Day Steering Committee. Obesity and kidney disease: hidden consequences of the epidemic. J Nephrol. 2017 Feb;30(1):1-10. doi: 10.1007/s40620-017-0377-y. PMID 28214961
- [Background] Kovesdy CP, Furth SL, Zoccali C. Obesity and kidney disease: hidden consequences of the epidemic. Braz J Med Biol Res. 2017 Apr 13;50(5):e6075. doi: 10.1590/1414-431X20166075. PMID 28423118
- [Background] Hassani V, Pazouki A, Nikoubakht N, Chaichian S, Sayarifard A, Shakib Khankandi A. The effect of gabapentin on reducing pain after laparoscopic gastric bypass surgery in patients with morbid obesity: a randomized clinical trial. Anesth Pain Med. 2015 Feb 1;5(1):e22372. doi: 10.5812/aapm.22372. eCollection 2015 Feb. PMID 25789237
- [Background] Rupniewska-Ladyko A, Malec-Milewska M, Kraszewska E, Pirozynski M. Gabapentin before laparoscopic sleeve gastrectomy reduces postoperative oxycodone consumption in obese patients: a randomized double-blind placebo-controlled trial. Minerva Anestesiol. 2018 May;84(5):565-571. doi: 10.23736/S0375-9393.17.12194-2. Epub 2017 Nov 6. PMID 29108405
- [Background] Zewinger S, Rauen T, Rudnicki M, Federico G, Wagner M, Triem S, Schunk SJ, Petrakis I, Schmit D, Wagenpfeil S, Heine GH, Mayer G, Floege J, Fliser D, Grone HJ, Speer T. Dickkopf-3 (DKK3) in Urine Identifies Patients with Short-Term Risk of eGFR Loss. J Am Soc Nephrol. 2018 Nov;29(11):2722-2733. doi: 10.1681/ASN.2018040405. Epub 2018 Oct 2. PMID 30279273
- [Background] Kim CS, Oak CY, Kim HY, Kang YU, Choi JS, Bae EH, Ma SK, Kweon SS, Kim SW. Incidence, predictive factors, and clinical outcomes of acute kidney injury after gastric surgery for gastric cancer. PLoS One. 2013 Dec 9;8(12):e82289. doi: 10.1371/journal.pone.0082289. eCollection 2013. PMID 24349249